CLINICAL TRIAL: NCT04717882
Title: Towards Medication Optimisation in the Last Phase of Life: iLIVE Medication Study
Brief Title: iLIVE Medication Study
Acronym: iLIVEmed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. dr. Stefan Sleijfer (Other)
Collaborators: Lund University (Other); Landspitali University Hospital (Other); Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. Stefan Sleijfer, Drs. E.E.C.M. Elsten (executive investigator), Prof. dr. C.C.D. van der Rijt (principal investigator), Prof. dr. Sleijfer (sponsor), Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NL72473.078.20
Record Dates: First submitted 2021-01-07; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Palliative Care
Keywords: Palliative care; Medication Therapy Management; Clinical Decision Support System (CDSS); Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Before-after study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients in the control arm will receive the usual treatment
- Intervention arm (Experimental): After crossing over to the intervention period, attending physicians will receive medication alerts from the Clinical Decision Support System (CDSS) within 1 week after inclusion of the patient. The medication alerts will be sent to the physician's email address. The physician is free to follow or ignore the advice in the alerts. If the physicians thinks these alerts are relevant for the patient, the physician will discuss these alerts with the patient and/or relatives. After this conversation, the physician will prescribe or deprescribe medications based on the alerts.
  Interventions: Device: CDSS-OPTIMED

INTERVENTIONS:
Device: CDSS-OPTIMED — The CDSS-OPTIMED is a software program that provides the physician with a personalized alert on whether to consider stopping or starting medication for a specific patient.
  Arms: Intervention arm

SUMMARY:
The iLIVE medication study is a before-after study where medication optimisation of patients with an estimated life expectancy of six months is investigated. The investigators will include 400 patients in 3 countries. The primary outcome is an assessment of the quality of life of patients, four weeks after baseline assessment

DETAILED DESCRIPTION:
Rationale: Patients in the last phase of life often use many medications until shortly before they die. This is partly inevitable, because these patients often experience multiple distressing symptoms. However, for a considerable number of medications currently often used at the end of life, the benefit is debatable, e.g. because they are aimed at the long-term prevention of illness.

Objective: the primary objective is to examine whether the use of a clinical decision support system (CDSS-OPTIMED), a personalized medication advice to attending physicians of patients in the last phase of life, contributes to patients' quality of life.

Main study endpoints: the primary outcome is an assessment of the quality of life of patients, four weeks after baseline assessment

Potential risks and benefits associated with participation: the intervention in the medication study supports physicians in using available evidence and knowledge when prescribing or deprescribing medication for patients in the last phase of life. The intervention does not involve experimental treatment or medication. The investigators expect no other risks than known side effects of (stopping) medications. The investigators are aware that the study population concerns vulnerable people who may experience fluctuating symptoms and levels of suffering across their disease trajectory. The investigators acknowledge the risk of overburdening participants. If patients feel burdened by participating in the study, they are encouraged to indicate that.

ELIGIBILITY:
Inclusion criteria for patients:

1. Patient is 18 years or over and provides informed consent to participate.
2. The patient is aware that recovering from his/her disease is unlikely, as assessed by the attending physician.
3. The patient agrees to participate in the iLIVE cohort study.
4. The attending physician would not be surprised if the patient would die within 6 months ('Surprise question').
5. If the physician is uncertain about the surprise question, the patient is eligible if presenting with at least one SPICT indicator. The SPICT™ is a tool to help professionals identify people with general indicators of poor or deteriorating health and clinical signs of life-limiting conditions for assessment and care planning, based on general or disease-specific indicators.

Inclusion criteria for relative/informal caregiver of included patients:

Relatives of included patients are asked to participate if they are: 18 years or over and provide informed consent to participate; aware that it is unlikely that the patient will recover from his/her disease; and capable of filling in a questionnaire in the country's main language or in English.

Exclusion Criteria:

1. The patient is incapable of filling in a questionnaire in the country's main language or in English (patients may be supported by relatives when filling in the questionnaire).
2. The attending physician makes the decision that the patient should not be included in the study due to e.g. illness burden, fast deterioration or imminent death, lack of trusting relationship with the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Patients' quality of life | 4 weeks after baseline assessment
  measured by the EORTC QLQ-C15-PAL QoL question

SECONDARY OUTCOMES:
Patients' symptoms | 4 weeks after baseline assessment
  measured by the ESAS
Use of medication of the patient | 4 weeks after baseline assessment
  measured by the medical file data and pharmacist's information system
Patient survival | From inclusion until death if patients die within the study period. If patient do not die within the study period, they will be followed up to a maximum of the full study period, i.e. a period of 2 years after start of the study
  measured by the time between inclusion until death
Satisfaction of the patient and relative with medication | 4 weeks after baseline assessment
  measured by the TSQM-9
Satisfaction of the attending physician with the CDSS-OPTIMED | 4 weeks after baseline assessment
  measured by a self-developed questionnaire
Episodes of symptomatic hypertension/hypotension/hyperglycaemia/hypoglycaemia and thrombo-embolic complications or bleeding events of the patient | If patients die within 6 months after inclusion, data will be collected retrospectively from baseline until death. If patients live longer than 6 months, data will be collected retrospectively from baseline until 6 months after baseline
  collected via medical file data, using a pre-structured checklist
Socio-demographic characteristics of the patient | Baseline
  Age, gender, current living situation, education, nationality, religion, socioeconomic status

OTHER OUTCOMES:
Development and training costs of the intervention | Retrospectively over full study period, i.e. a period of 2 years
  Based on proformas completed by the developers and the study personnel
Operational costs of the intervention | Retrospectively over full study period, i.e. a period of 2 years
  Based on time spent on discussing medication alerts with the pharmacist and patient/relative and time registrations via automated system extracts
Patients' use of medical interventions | If patients die within 6 months after inclusion, data will be collected retrospectively from baseline until death. If patients live longer than 6 months, data will be collected retrospectively from baseline until 6 months after baseline
  Measured by using a pre-structured checklist. Items to be assessed include: place of care, medical events and complications, medication use, medical and surgical interventions, goals of care statements, resuscitation policy, non-treatment decisions
Costs of medical care | If patients die within 6 months after inclusion, data will be collected retrospectively from baseline until death. If patients live longer than 6 months, data will be collected retrospectively from baseline until 6 months after baseline
  Measured by using a pre-structured checklist. Items to be assessed include: place of care, medical events and complications, medication use, medical and surgical interventions, goals of care statements, resuscitation policy, non-treatment decisions
Patients' health related quality of life | 4 weeks after baseline assessment
  measured by the EQ-5D-5L
Patients' capabilities | 4 weeks after baseline assessment
  measured by the ICECAP-SCM
Patients' resource use, employment and patient activities/informal care needs | 4 weeks after baseline assessment
  measured by the HEQ
Relatives' health related quality of life | 4 weeks after baseline assessment
  measured by the EQ-5D-5L
Relatives' capabilities | 4 weeks after baseline assessment
  measured by the ICECAP-CPM
Relatives' informal care provision | 4 weeks after baseline assessment
  measured by the partial IVICQ and CIIQ
Dutch subgroup patients' health related quality of life | 8 weeks after baseline assessment, repeated 4-weekly to a maximum of 24 weeks
  measured by the EQ-5D-5L
Dutch patients' capabilities | 8 weeks after baseline assessment, repeated 4-weekly to a maximum of 24 weeks
  measured by the ICECAP-SCM
Dutch patients' resource use, employment and patient activities/informal care needs | 8 weeks after baseline assessment, repeated 4-weekly to a maximum of 24 weeks
  measured by the HEQ

CONTACTS AND LOCATIONS:
Overall Officials: Karin van der Rijt, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Erasmus Medical Center, Rotterdam, Netherlands
- Skåne University Hospital, Lund, Sweden
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes